CLINICAL TRIAL: NCT01119846
Title: A Study in Type II Diabetic Subjects of Single and Multiple Doses of Orally Administered GSK1292263 to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Compound Alone and When Co-administered With Sitagliptin or Metformin
Brief Title: A Study in Type 2 Diabetics of Single and Multiple Doses of Orally Administered GSK1292263 to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 111598
Record Dates: First submitted 2009-11-12; First posted 2010-05-10 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Tolerability; Pharmacokinetics; Safety; Pharmacodynamics; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (1-(3-isopropyl-1,2,4-oxadiazol-5-yl)piperidin-4-yl)methyl methanesulfonate; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): Part A (Cohort 1) is a single-blind, randomized, placebo-controlled, 5-period crossover in which drug naïve T2DM subjects will receive escalating doses of GSK1292263 in each of 3 periods and placebo and open-label sitagliptin in the other 2 periods. The sequence will be randomized, but will maintain the low, medium and high dose order for GSK1292263.
  Interventions: Drug: GSK1292263; Drug: GSK1292263 matching placebo; Drug: Sitagliptin
- Part B (Experimental): Part B (Cohort 2) is a single-blind, randomized, 2-period study in which T2DM subjects will receive a single dose of GSK1292263, fasted or fed.
  Interventions: Drug: GSK1292263
- Part C (Experimental): Part C (Cohort 3, optional Cohort 4) is a single-blind, randomized, placebo-controlled, 5-arm study of 14 days of dosing with GSK1292263, placebo or open-label sitagliptin. An optional Cohort 4 may be enrolled to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK1292263 when dosed in a BID regimen.
  Interventions: Drug: GSK1292263; Drug: GSK1292263 matching placebo; Drug: Sitagliptin

INTERVENTIONS:
Drug: GSK1292263 — GSK1292263 is an immediate-release round, white, film-coated tablet provided in 3 strengths, 25mg, 75mg and 200mg being developed for the treatment of type 2 diabetes.
Drug: GSK1292263 matching placebo — Matching placebo to active drug GSK1292263
  Arms: Part A; Part C
Drug: Sitagliptin — Sitagliptin (Januvia) 100mg tablets are beige, round, film-coated tablets with "277" on one side.
  Other Names: Januvia
  Arms: Part A; Part C

SUMMARY:
The purpose of this study is to see if GSK1292263 is safe and well-tolerated when administered to type 2 diabetics, and to get preliminary information about whether it may be effective in the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
Data from this study will be used to assess the potential of GSK1292263 as a treatment for T2DM, and will aid the design and dose selection of future studies of longer duration in T2DM subjects that will evaluate GSK1292263 alone or in combination with other anti-diabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 - 60 years of age, inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. FSH and estradiol levels will be checked at Screening for postmenopausal women. Simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40pg/ml (<140pmol/L) is confirmatory.
* Except as noted elsewhere, subjects should have no significant known medical conditions other than T2DM, as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECGs. A subject with a clinical abnormality or laboratory parameters that meets exclusion criteria but is outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* BMI (body mass index) within the range 22-35 kg/m2, inclusive.
* Part A - T2DM diagnosed by American Diabetes Association criteria at least 3 months prior to Screening with:
* Currently controlled by diet and exercise.
* Fasting plasma glucose (FPG) level <= 250mg/dL at the Screening visit
* FPG level <= 250mg/dL on Day -1
* HbA1c between 6.5 and 11%, inclusive, at Screening visit
* For Parts B and C, T2DM diagnosed by American Diabetes Association criteria at least 3 months prior to Screening with:
* T2DM currently controlled by diet and exercise, or, if on medication, subjects must be treating their T2DM using one of the following regimens:
* Metformin as monotherapy
* Sulfonylurea as monotherapy
* Metformin and sulfonylurea in combination, if both components are being administered at doses that are half their maximum dose or less
* DPP-IV inhibitors, either as monotherapy or in combination with other agent(s) on this list at half maximal dose or less
* Exenatide, either as monotherapy or in combination with other agent(s) on this list at half maximal dose or less
* For subjects that are being screened for Parts B and C, all doses of anti-diabetic medication must have been stable for at least 3 months prior to Screening, and the subject must be willing to wash out from their anti-diabetic medications from Day -7 through post-last-dose of Period 2 (Part B) or Day -7 through Day 15 (Part C).
* Fasting plasma glucose (FPG) level <= 220mg/dL at the Screening visit
* FPG level <= 250mg/dL on Day -1
* HbA1c between 7 and 11%, inclusive, at Screening visit
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Has any of the following laboratory abnormalities:
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C, result within 3 months of screening.
* Positive test for HIV antibody.
* History of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by TSH at Screening. (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy for at least 3 months prior to Screening and who have a screening thyroid stimulating hormone (TSH) within the normal range may participate.)
* ALT and/or AST > 2 times the upper limit of normal at screening.
* Fasting triglycerides > 450mg/dL at screening.
* Total Bilirubin > 1.5 times the upper limit of normal at screening.
* For females a haemoglobin < 11.5 g/dL, and for males a hemoglobin < 12.5 g/dL. Hemoglobin < 11g/dL(A female subject with haemoglobin between 10g/dL and 11.5 g/dL, or a male subject with haemoglobin between 10g/dL and 12.5 g/dLmay be enrolled only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk to the subject and will not interfere with the study procedures).
* A positive pre-study drug/urine screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A pre-study urine cotinine screen indicating use of tobacco/ nicotine containing products.
* If female is pregnant or has a positive pregnancy test
* Significant renal disease as manifested by one or more of the following:
* Creatinine clearance <60mL/min. (estimated from serum creatinine (SCr) and demographic data using the MDRD calculation):
* To calculate estimated GFR (mL/min/1.73m2) manually:

=186 x (SCr in mg/dL)-1.154 x (age)-0.203 x (0.742 if female) x (1.210 if African-American) =exp (5.228-1.154 x ln (SCr)-0.203x ln(age)-(0.299 if female) + (0.192 if African American)) (A link to a validated MDRD calculator on the internet is provided in the SRM.)

* Urine protein/creatinine (mg of protein/mg of creatinine) ratio >2.5; or urine albumin concentration >300mg/g of creatinine).
* Known loss of a kidney either by surgical ablation, injury, or disease.
* Significant ECG abnormalities, defined as follows:

Heart Rate < 50 and >100bpm PR Interval <120 and > 220ms QRS duration < 70 and >120ms QTC Interval (Bazett)* > 450ms

Or, has clinically significant rhythm abnormalities identified during 24-hour Screening Holter assessment. Subjects with Left Bundle Branch Block are excluded from the study. Subjects with partial Right Bundle Branch Block may be considered for inclusion following consultation with the GSK Medical Monitor. Subjects with WPW syndrome are excluded from the study.

*Note that if ECG abnormalities are identified, the ECG should be repeated two more times (with 5 minutes between ECG readings) and the average of the 3 values used to determine eligibility.

* Systolic pressure > 150mmHg or <80mmHg or diastolic blood pressure > 95mmHg or <60mmHg at screening. Blood pressure assessments may be repeated once if needed, allowing adequate time for subject to rest.
* Previous use of insulin as a treatment within 3 months of Screening, or for >2 weeks when used for acute illness in the last 12 months prior to Screening, or if used for more than 1 year when associated with gestational diabetes mellitus.
* Has a history of any of the following conditions:
* Clinically significant symptoms of gastroparesis
* Cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to Screening
* Gastrointestinal disease that could affect fat or bile acid absorption, including inflammatory bowel disease, chronic diarrhea, Crohn's or malabsorption syndromes within the past year
* Gastrointestinal surgery
* Chronic or acute pancreatitis
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360mL) of beer, 5 ounces (150mL) of wine or 1.5 ounces (45mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Is taking prohibited medications. See Section 9.3 for a detailed list of prohibited medications. Note also:
* The use of anti-diabetic agents other than those listed in Inclusion #7 is reason for exclusion and subjects will not be allowed to wash off of unapproved anti-diabetic medications in order to qualify for participation in this study.
* Subjects must wash out from the following medications during the 7-day period prior to first dose, and must remain off these medications through discharge on post-last-dose of Period 2 (Part B) or Day 15 (Part C): all anti-diabetic medications specified in Inclusion #7, all statin agents, fat absorption blocking agents, bile acid sequestrants. Fibrates must be washed out for a 14-day period prior to first dose.
* Vitamins, herbal and dietary supplements (including St John's Wort) are prohibited within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication and through discharge.
* Unwilling to abstain from
* Caffeine-or xanthine-containing products for 24 hours prior to dosing until post-last-dose of Period 5 (Part A), post-last-dose of Period 2 (Part B) or Day -7 through Day 15 (Part C).
* Use of illicit drugs or nicotine-containing products
* Alcohol for 24 hours prior to dosing until post-last-dose of Period 5 (Part A), post-last-dose of Period 2 (Part B) or Day -7 through Day 15 (Part C).
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic blood samples.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. This includes sensitivity to heparin or heparin-induced thrombocytopenia, if heparin will be used to maintain catheter patency.
* Where participation in the study would result in donation of blood in excess of approximately 500mL within a 56 day period.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06-05 (Actual); Primary Completion 2010-03-19 (Actual); Study Completion 2010-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Nunez DJ, Bush MA, Collins DA, McMullen SL, Gillmor D, Apseloff G, Atiee G, Corsino L, Morrow L, Feldman PL. Gut hormone pharmacology of a novel GPR119 agonist (GSK1292263), metformin, and sitagliptin in type 2 diabetes mellitus: results from two randomized studies. PLoS One. 2014 Apr 3;9(4):e92494. doi: 10.1371/journal.pone.0092494. eCollection 2014. PMID 24699248
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111598 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13, 4 and 83 participants with type 2 diabetes mellitus (T2DM) were randomized in Part A, B and C, respectively. The study was conducted from 05 June 2009 to 19 March 2010 at 8 centers in the United States.
Pre-assignment Details: The maximum time a participant spent in Part A, B and C of the study was approximately 10, 7 and 7 weeks, respectively including the 28-days period allotted for screening assessments in all parts.
Groups:
- Part A: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive escalating doses of GSK1292263 25 milligrams (mg), 150 mg and 800 mg in each of 3 periods along with placebo and sitagliptin 100 mg orally in the other 2 periods in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the oral glucose tolerance test (OGTT).
- Part B: In this part (Cohort 2), after the appropriate washout period, T2DM participants on monotherapy or sub-maximal anti-diabetic medications were randomized to receive a single dose of GSK1292263 800 mg orally in fasted or fed condition. Before participants in Part B were dosed, the safety and tolerability of GSK1292263 800 mg administered in the fasted state to 9 participants in Part A was reviewed to ensure that it was safe to proceed. In Part B, study drug was administered 30 minutes after breakfast and lunch and dinner was approximately 4 and 10 hours after dosing.
- Part C: Participants were randomized to 14 days of dosing with 4 dose regimens of GSK1292263 (final doses were: 50 mg twice daily [BID], 150 mg BID, 300 mg BID, and 600 mg once daily) or matching placebo (administered BID) or open-label sitagliptin 100 mg (dosed once daily with the morning dose of GSK1292263). In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
Period: Overall Study
Arm/Group | Part A | Part B | Part C
Started | 13 | 4 | 83
Completed | 11 | 4 | 72
Not Completed | 2 | 0 | 11
Not completed — Adverse Event | 1 | 0 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Part A: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive escalating doses of GSK1292263 25 mg, 150 mg and 800 mg in each of 3 periods along with placebo and sitagliptin 100 mg orally in the other 2 periods in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part B: In this part (Cohort 2), eligible T2DM participants on mono-therapy or sub-maximal anti-diabetic medications washed off these medications for 1 week and received a single dose of GSK1292263 800 mg orally in fasted or fed condition. Before participants in Part B were dosed, the safety and tolerability of GSK1292263 800 mg administered in the fasted state to 9 participants in Part A was reviewed to ensure that it was safe to proceed. In Part B, study drug was administered 30 minutes (min) after breakfast and lunch and dinner was approximately 4 and 10 hours after dosing.
- Part C: Participants were randomized to 14 days of dosing with 4 dose regimens of GSK1292263 (final doses were: 50 mg BID, 150 mg BID, 300 mg BID, and 600 mg once daily) or matching placebo (administered BID) or open-label sitagliptin 100 mg (dosed once daily with the morning dose of GSK1292263). In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa.
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Part C | Total
Number analyzed (Participants) | 13 | 4 | 83 | 100
Age, Customized [Count of Participants; unit: Participants]
  18-60 Years | 13 | 4 | 83 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 22 | 27
  Male | 9 | 3 | 61 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 6 | 8
  White | 12 | 3 | 75 | 90
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to Week 10
Population: Safety Population comprised of all participants enrolled in the study and who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive placebo orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: GSK1292263 25 mg: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive GSK1292263 25 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: GSK1292263 150 mg: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive GSK1292263 150 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: GSK1292263 800 mg: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive GSK1292263 800 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: Sitagliptin 100 mg: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive sitagliptin 100 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Participants
  Any AE | 2 | 2 | 2 | 4 | 2
  Any SAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants With Abnormal Hematology Parameters of Potential Clinical Importance (PCI)
Description: Hematology parameters included platelet count, red blood cell (RBC) count, mean corpuscular volume (MCV), total neutrophils, white blood cell count (WBC; absolute), mean corpuscular hemoglobin (MCH), lymphocytes, mean corpuscular hemoglobin concentration (MCHC), monocytes, hemoglobin, eosinophils, hematocrit, reticulocytes and basophils. It was assessed on Screening, Day -1, Day 2 (of each treatment period) and Follow-up (7 to 10 days after final discharge). Only those parameters (hemoglobin, high) for which at least one value of PCI was reported are summarized. Null data is not presented.
Time Frame: Up to Week 10
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Participants | 0 | 0 | 1 | 0 | 1

3. Primary Outcome: Part A: Number of Participants With Abnormal Clinical Chemistry Parameters of PCI
Description: Clinical chemistry parameters included blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), total and direct bilirubin, creatinine, chloride, alanine aminotransferase (ALT), uric acid, glucose fasting, gamma glutamyltransferase (GGT), albumin, sodium, magnesium, phosphorus inorganic, calcium, total carbon dioxide (CO2), alkaline phosphatase (ALP), triglycerides, total cholesterol, low-density lipoprotein (LDL) cholesterol, free fatty acid (non-esterified fatty acids; [NEFA]), high-density lipoprotein (HDL) cholesterol and total protein. It was assessed on Screening, Day -1, Day 2 (of each treatment period) and Follow-up (7 to 10 days after final discharge). Only those parameters for which at least one value of PCI was reported are summarized. Null data is not presented.
Time Frame: Up to Week 10
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Participants
  Glucose, High | 0 | 1 | 0 | 0 | 0
  CO2, Low | 0 | 1 | 0 | 0 | 0
  Magnesium, High | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Part A: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs was obtained in a supine position at each time point during the study using an ECG machine that automatically measured PR, QRS, QT and QTc intervals (QT duration corrected for heart rate by Bazett's formula [QTcB] and Fridericia's formula [QTcF]). Participants with abnormal clinically significant ECG findings is presented. It was assessed on Screening, Day 1 at pre-dose, 1, 2, 3, 4, 6, 10, 16, 24 hours and Follow-up (7 to 10 days after final discharge).
Time Frame: Up to Week 10
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Abnormal Vital Signs of PCI
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate measurements were recorded at each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes. Participants with abnormal clinically significant vital signs findings is presented. It was assessed on Screening, Day -1, 1, 2 (pre-dose, 1, 3, 4, 6, 10, 16 and 24 hours of each treatment period) and Follow-up (7 to10 days after final discharge).
Time Frame: Up to Week 10.
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part A: Summary of Maximum Plasma Concentration (Cmax)
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. Blood samples for the determination of PKs was collected at on Day 1 of each period: immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 14 and 24 hours.
Time Frame: Pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 14 and 24 hours on Day 1 of each treatment period
Population: The Pharmacokinetic Population included all participants from the Safety Population who have any pharmacokinetic parameter estimates from any portion of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliters
Arm/Group | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg
Number analyzed (Participants) | 12 | 12 | 11
Nanograms per milliliters | 52.04 (17.147) | 165.62 (37.467) | 379.79 (28.171)
Statistical Analysis 1: Comparison: Part A: GSK1292263 25 mg vs Part A: GSK1292263 150 mg vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Slope = 0.5782, 90% CI 2-sided [0.5230 to 0.6335] — Dose Proportionality for GSK1292263 Using the Power Model

7. Primary Outcome: Part A: Summary of Time to Maximum Concentration (T-max) and Lag Time Before Observation of Drug Concentration in Sampled Matrix (T-lag)
Description: The time at which Cmax was observed was determined directly from the raw concentration-time data. The lag time before observation of drug concentrations in sample matrix determined as the time of the sample preceding the first quantifiable concentration. Blood samples for the determination of PK was collected on Day 1 of each period: immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 14 and 24 hours.
Time Frame: Pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 14 and 24 hours on Day 1 of each treatment period
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg
Number analyzed (Participants) | 12 | 12 | 11
Hour
  T-lag | 0.50 [0.0 to 1.0] | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.5]
  T-max | 4.99 [1.0 to 6.0] | 3.00 [2.0 to 8.0] | 3.00 [1.9 to 6.0]

8. Primary Outcome: Part A: Summary of Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC0-t) and Area Under the Concentration-time Curve From Zero (Pre-dose) to 24 Hours (AUC0-24)
Description: The AUC 0-24 and AUC 0-t determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples for the determination of PK was collected at on Day 1 of each period: immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 14 and 24 hours.
Time Frame: Pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 14 and 24 hours on Day 1 of each treatment period
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms×hour per milliliters
Arm/Group | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg
Number analyzed (Participants) | 12 | 12 | 11
Nanograms×hour per milliliters
  AUC 0-24 | 524.30 (21.138) | 1684.86 (31.009) | 3985.72 (28.449)
  AUC 0-t | 526.88 (20.208) | 1685.44 (31.015) | 3979.35 (27.457)
Statistical Analysis 1: Comparison: Part A: GSK1292263 25 mg vs Part A: GSK1292263 150 mg vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Slope = 0.5828, 90% CI 2-sided [0.5282 to 0.6375] — Dose Proportionality for GSK1292263 Using the Power Model for AUC0-24
Statistical Analysis 2: Comparison: Part A: GSK1292263 25 mg vs Part A: GSK1292263 150 mg vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Slope = 0.5808, 90% CI 2-sided [0.5325 to 0.6291] — Dose Proportionality for GSK1292263 Using the Power Model for AUC0-last

9. Primary Outcome: Part C: Number of Participants With AEs and SAEs
Description: An AE was defined as any untoward MO in a participant temporally associated with the use of a MP, whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: GSK1292263 50 mg BID: Participants were randomized to 14 days of dosing with GSK1292263 50 mg BID once daily. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: GSK1292263 150 mg BID: Participants were randomized to 14 days of dosing with GSK1292263 150 mg BID once daily. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: GSK1292263 300 mg BID: Participants were randomized to 14 days of dosing GSK1292263 300 mg BID. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: GSK1292263 600 mg Once Daily: Participants were randomized to 14 days of dosing GSK1292263 600 mg once daily. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: Placebo: Participants were randomized to 14 days of dosing with matching placebo (administered BID). In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: Sitagliptin 100 mg: Participants were randomized to 14 days of dosing with open-label sitagliptin 100 mg (dosed once daily with the morning dose of GSK1292263). In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 16 | 12 | 14 | 15 | 12
Participants
  Any AE | 4 | 5 | 1 | 4 | 4 | 2
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part C: Number of Participants With Abnormal Hematology Parameters of PCI
Description: Hematology parameters included platelet count, RBC count, MCV, total neutrophils, WBC absolute, MCH, lymphocytes, MCHC, monocytes, hemoglobin, eosinophils, hematocrit, reticulocytes and basophils. It was assessed on Screening, Day -2 (can be non-fasting) and prior to breakfast (early in the morning, fasting) on Days 1, 7 and 14, and on Day 15 prior to checkout, (=24 hours post-dose) of each treatment period and Follow-up (7 to 10 days after final discharge). Only those parameters for which at least one value of PCI was reported are summarized. Null data is not presented.
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 16 | 12 | 14 | 15 | 12
Participants
  Hematocrit, High | 0 | 0 | 0 | 1 | 0 | 0
  Hemoglobin, High | 0 | 0 | 0 | 2 | 0 | 2
  Total neutrophils, Low | 0 | 0 | 0 | 2 | 0 | 1

11. Primary Outcome: Part C: Number of Participants With Abnormal Clinical Chemistry Parameters of PCI
Description: Clinical chemistry parameters included BUN, potassium, AST, total and direct bilirubin, creatinine, chloride, ALT, uric acid, glucose fasting, GGT, albumin, sodium, magnesium, phosphorus inorganic, calcium, total CO2, ALP, triglycerides, total cholesterol, LDL cholesterol, free fatty acid (NEFA), HDL cholesterol and total protein. It was assessed on Screening, Day -2 (can be non-fasting) and prior to breakfast (early in the morning, fasting) on Days 1, 7 and 14, and on Day 15 prior to checkout, (=24 hours post-dose) of each treatment period and Follow-up (7 to 10 days after final discharge). Only those parameters for which at least one value of PCI was reported are summarized. Null data is not presented.
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 15 | 12 | 14 | 16 | 12
Participants
  Phosphorus inorganic, Low | 0 | 0 | 0 | 0 | 1 | 0
  CO2, High | 1 | 0 | 0 | 0 | 1 | 1
  Glucose, High | 5 | 1 | 4 | 4 | 3 | 3
  CO2, Low | 0 | 0 | 0 | 0 | 1 | 0
  Potassium, Low | 0 | 0 | 0 | 0 | 1 | 0
  ALT, High | 0 | 0 | 0 | 0 | 1 | 0
  Albumin, Low | 1 | 0 | 0 | 0 | 0 | 0
  Calcium, Low | 1 | 0 | 0 | 0 | 0 | 0
  Sodium, Low | 0 | 1 | 0 | 0 | 0 | 0

12. Primary Outcome: Part C: Number of Participants With Significant ECG Abnormalities
Description: Twelve-lead ECGs was obtained in a supine position at each time point during the study using an ECG machine that automatically measured PR, QRS, QT and QTc intervals (QTcB and QTcF). Participants with abnormal clinically significant ECG findings is presented. It was assessed on Screening, on Day -1, 1, 7, 13 and 14 pre-breakfast dose (fasting) and at 1, 3, 6, 9, 12 and 24 hours of each treatment period and Follow-up (7 to 10 days after final discharge).
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 15 | 12 | 14 | 16 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Part C: Number of Participants With Abnormal Vital Signs of PCI
Description: SBP, DBP and pulse rate measurements were recorded at each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes. Participants with abnormal clinically significant vital signs findings is presented. It was assessed on Screening, on Days -1 to 14 in a fasting state early in the morning (prior to morning dosing on days 1-14) and at Follow-up. On Days 1, 7, 13 and 14, it was also taken at 1, 3, 6, 9, 12 and 24 hours after the morning dose each treatment period and Follow-up (7 to 10 days after final discharge).
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 15 | 12 | 14 | 16 | 12
Participants
  SBP, Low | 0 | 0 | 0 | 1 | 0 | 0
  SBP, High | 0 | 0 | 1 | 0 | 2 | 0
  Pulse rate, High | 0 | 0 | 0 | 1 | 0 | 0

14. Primary Outcome: Part C: Summary of Plasma Cmax
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (= post-breakfast), 1, 2, 4 (= pre-lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: Pharmacokinetic Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Nanograms per millimeter
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily
Number analyzed (Participants) | 14 | 15 | 12 | 13
Nanograms per millimeter
  Day 1 | 219.36 (14.140) | 364.73 (29.202) | 584.32 (30.096) | 721.18 (23.346)
  Day 7: number analyzed (Participants) | 12 | 15 | 12 | 12
  Day 7 | 410.98 (25.083) | 715.01 (26.989) | 1149.32 (25.481) | 813.03 (24.578)
  Day 13: number analyzed (Participants) | 12 | 12 | 11 | 11
  Day 13 | 433.12 (20.372) | 732.05 (29.116) | 969.19 (31.059) | 831.23 (18.373)
  Day 14: number analyzed (Participants) | 12 | 12 | 11 | 11
  Day 14 | 438.36 (19.487) | 715.71 (30.769) | 950.52 (35.046) | 772.89 (23.019)

15. Primary Outcome: Part C: Summary of T-max and T-lag
Description: The time at which Cmax was observed was determined directly from the raw concentration-time data. The lag time before observation of drug concentrations in sample matrix determined as the time of the sample preceding the first quantifiable concentration. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (= post-breakfast), 1, 2, 4 (= pre-lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: Pharmacokinetic Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily
Number analyzed (Participants) | 14 | 15 | 12 | 13
Hour
  T-lag, Day 1 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.50 [0.0 to 0.5]
  T-max, Day 1 | 4.00 [4.0 to 12.0] | 12.00 [2.0 to 12.0] | 12.00 [2.0 to 12.0] | 3.97 [1.50 to 14.0]
  T-max, Day 7: number analyzed (Participants) | 12 | 15 | 12 | 12
  T-max, Day 7 | 3.97 [2.0 to 12.0] | 3.97 [0.0 to 12.0] | 3.97 [0.0 to 12.0] | 4.0 [4.0 to 6.0]
  T-max, Day 13: number analyzed (Participants) | 12 | 12 | 11 | 11
  T-max, Day 13 | 3.97 [2.0 to 12.0] | 3.98 [2.0 to 12.0] | 3.97 [0.0 to 12.0] | 3.97 [2.0 to 6.0]
  T-max, Day 14 | 4.01 [4.0 to 12.0] | 3.98 [1.0 to 6.0] | 3.98 [1.0 to 12.0] | 3.98 [3.9 to 4.0]

16. Primary Outcome: Part C: Summary of AUC0-10, AUC0-12 and AUC0-24
Description: The AUC0-10, AUC0-12 and AUC0-24 determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For QD and BID dosing regimens on Day 7, blood samples were collected at pre-dose (=post- breakfast), 1, 2, 4 (=pre lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily
Number analyzed (Participants) | 14 | 15 | 12 | 13
Ratio
  AUC 0-10, Day 1 | 1127.45 (10.341) | 1868.87 (24.974) | 3076.52 (23.023) | 4003.80 (27.722)
  AUC 0-10, Day 13: number analyzed (Participants) | 12 | 12 | 11 | 11
  AUC 0-10, Day 13 | 3167.19 (21.745) | 5869.82 (32.289) | 7332.26 (32.746) | 5348.21 (22.627)
  AUC 0-10, Day 14: number analyzed (Participants) | 12 | 12 | 11 | 11
  AUC 0-10, Day 14 | 3179.51 (22.197) | 5723.55 (32.728) | 7451.13 (37.067) | 5470.57 (23.708)
  AUC 0-12, Day 7: number analyzed (Participants) | 12 | 15 | 12 | 12
  AUC 0-12, Day 7 | 3559.59 (27.687) | 6413.05 (31.719) | 9965.14 (27.260) | 6268.95 (27.159)
  AUC 0-24, Day 1 | 3552.46 (15.595) | 6439.56 (26.152) | 11078.97 (24.411) | 7153.16 (34.663)
  AUC 0-24, Day 13: number analyzed (Participants) | 12 | 12 | 11 | 11
  AUC 0-24, Day 13 | 7776.26 (23.727) | 14463.50 (29.668) | 18682.34 (32.153) | 9388.93 (26.616)
  AUC 0-24, Day 14: number analyzed (Participants) | 12 | 12 | 11 | 11
  AUC 0-24, Day 14 | 8026.26 (22.275) | 14356.75 (29.796) | 19134.61 (34.542) | 10166.83 (26.747)

17. Primary Outcome: Part C: Summary of Accumulation Ratio (Ro)
Description: Ro was derived as follows: Ro = Day 13 (AUC0-24)/Day 1 (AUC0-24) for once daily dosing; Ro = Day 13 AM (AUC0-10)/Day 1 AM (AUC0-10) for BID dosing and Ro = Day 13 (AUC0-24)/Day 1 (AUC0-24) for BID dosing. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (= post-breakfast), 1, 2, 4 (= pre-lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected. Data presented for Day 13 and Day 14.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily
Number analyzed (Participants) | 14 | 15 | 12 | 13
Ratio
  Day 13: number analyzed (Participants) | 12 | 12 | 11 | 11
  Day 13 | 2.22 (21.131) | 2.17 (19.972) | 1.72 (31.647) | 1.29 (40.690)
  Day 14: number analyzed (Participants) | 12 | 12 | 11 | 11
  Day 14 | 2.29 (19.681) | 2.15 (20.319) | 1.77 (31.510) | 1.39 (39.448)

18. Primary Outcome: Part C: Summary of Time Invariance Ratio (Rs) of AUC0-10 for BID Dose of GSK1292263
Description: The AUC0-10 determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (=post-breakfast), 1, 2, 4 (=pre lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID
Number analyzed (Participants) | 14 | 15 | 12
Ratio | 2.8174 [2.5262 to 3.1422] | 3.0033 [2.6743 to 3.3727] | 2.4218 [2.0455 to 2.8673]

19. Primary Outcome: Part C: Summary of Time Invariance Ratio (Rs) of AUC0-24 for Once Daily Dose of GSK1292263
Description: The AUC0-24 determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (=post-breakfast), 1, 2, 4 (=pre lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part C: GSK1292263 600 mg Once Daily
Number analyzed (Participants) | 11
Ratio | 1.2871 [1.0392 to 1.5941]

20. Primary Outcome: Part C: Summary of Time Invariance Ratio (Rs) of Cmax
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (=post-breakfast), 1, 2, 4 (=pre lunch), 6, 10 (=immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected. Cmax for one participant from 50 BID x 14 day was not analyzed due to positive definite G Matrix.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily
Number analyzed (Participants) | 15 | 12 | 13
Ratio | 1.9186 [1.6979 to 2.1680] | 1.6755 [1.4769 to 1.9007] | 1.1703 [1.0414 to 1.3152]

21. Primary Outcome: Part A: Relationships Between GSK1292263 Drug Exposures and Insulin Sensitivity
Description: Blood samples for the determination of insulin were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. For lunch and evening meal in Part A, samples were collected just before the meal and at the following times after starting each meal: 0.5, 1, 1.5 (except breakfast in Part B), 2 and 3 hours. When this results in multiple samples at the same time point, only one sample was collected. The unit of measure is mL/min×1/micro international unit×10^4 (mL/min×1/µIU×10^4).
Time Frame: Day 1 of each treatment period
Population: The PK/PD Population included all participants who were in both the PK and PD populations, as well as those in the PD population who received the placebo treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min×1/µIU×10^4
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 12
mL/min×1/µIU×10^4 | 1.4 (98) | 2.1 (67) | 2.3 (51) | 2.8 (86) | 2.7 (86)

22. Primary Outcome: Part C: Relationships Between GSK1292263 Drug Exposures and Insulin Sensitivity
Description: Blood samples for the determination of insulin were collected fasting pre-breakfast and then pre-morning dose (PD time 0) on Days -1, 13 and 14, and then at 10, 20, 30, 60, 90, 120, 180 min after eating the standardized breakfast meal tolerance test. For lunch (approximately 4 hour post-morning dose) samples were collected just before the meal and at the following times after starting each meal: 0.5, 1, 1.5, 2 and 3 hours. For the evening meal (approximately 10 hour post-morning dose), BID dosing groups followed the sequence of sampling, food and dosing as for breakfast (PD sample immediately before meal, eat and then dose), then 0.5, 1, 1.5, 2 and 3 hours post-dinner. A sample was also collected 24 hours post-dose.
  When this results in multiple samples at the same time point, only one sample was collected (example: 24 hours post first-dose = pre-dose [time 0] for the second dose).
Time Frame: Day -1, 13 and 14
Population: PK/PD Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min×1/µIU×10^4
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
mL/min×1/µIU×10^4
  Day -1: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 12
  Day -1 | 6.4 (149) | 9.8 (100) | 9.2 (80) | 8.0 (96) | 6.6 (79) | 7.0 (107)
  Day 13: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 11
  Day 13 | 5.6 (64) | 8.6 (50) | 8.7 (99) | 7.2 (72) | 6.6 (59) | 7.4 (122)
  Day 14: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 11
  Day 14 | 5.7 (88) | 9.0 (52) | 7.3 (90) | 8.0 (75) | 6.8 (91) | 5.7 (124)

23. Primary Outcome: Part A: Summary of Change From Baseline in Fasted Glucose
Description: Blood samples for the determination of glucose were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. For lunch and evening meal in Part A, samples were collected just before the meal and at the following times after starting each meal: 0.5, 1, 1.5 (except breakfast in Part B), 2 and 3 hours. When this results in multiple samples at the same time point, only one sample was collected. Change from Baseline was calculated by subtracting Baseline value from post-Baseline value. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Baseline (Day 1 pre-dose) and Day 1 (24 hours)
Population: The PD Population included participants from the Safety Population who had any PD parameter estimates from any portion of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millimoles per Liter
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Millimoles per Liter | 0.52 (795.822) | 1.49 (848.906) | 0.53 (533.024) | 0.87 (653.005) | 0.58 (-220.270)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.036, 95% CI 2-sided [-1.17 to 1.10]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Net) = 0.225, 95% CI 2-sided [-0.90 to 1.35]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Net) = 0.046, 95% CI 2-sided [-1.10 to 1.19]
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.679, 95% CI 2-sided [-1.80 to 0.45]

24. Primary Outcome: Part A: Summary of the AUC 0-13, AUC 0-24, Incremental AUC (iAUC) 0-13 and iAUC 0-24 of Glucose
Description: Blood samples for the determination of glucose were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. For lunch and evening meal in Part A, samples were collected just before the meal and at the following times after starting each meal: 0.5, 1, 1.5 (except breakfast in Part B), 2 and 3 hours. When this results in multiple samples at the same time point, only one sample was collected. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millimoles per Liter
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Millimoles per Liter
  AUC 0-13 | 9.42 (16.011) | 9.44 (24.357) | 9.15 (21.389) | 8.64 (20.241) | 9.23 (39.431)
  AUC 0-24: number analyzed (Participants) | 10 | 12 | 12 | 11 | 13
  AUC 0-24 | 8.72 (17.563) | 9.17 (22.684) | 9.03 (20.928) | 8.67 (18.128) | 8.95 (33.715)
  iAUC 0-13 | 2.11 (32.518) | 1.35 (62.815) | 1.48 (59.021) | 1.78 (64.653) | 1.48 (97.908)
  iAUC 0-24: number analyzed (Participants) | 10 | 12 | 12 | 11 | 13
  iAUC 0-24 | 1.18 (43.037) | 1.04 (96.395) | 1.44 (137.548) | 0.90 (141.078) | 0.53 (188.368)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.265, 95% CI 2-sided [-1.80 to 2.33] — Comparison of AUC(0-24)
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.614, 95% CI 2-sided [-1.53 to 2.76] — Comparison of AUC(0-24)
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.451, 95% CI 2-sided [-1.64 to 2.54] — Comparison of AUC(0-24)
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.469, 95% CI 2-sided [-1.39 to 2.33] — Comparison of AUC(0-24)
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.290, 95% CI 2-sided [-2.53 to 1.95] — Comparison of AUC(0-13)
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-2.35 to 2.30] — Comparison of AUC(0-13)
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.163, 95% CI 2-sided [-2.48 to 2.15] — Comparison of AUC(0-13)
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.167, 95% CI 2-sided [-1.88 to 2.21] — Comparison of AUC(0-13)
Statistical Analysis 9: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.352, 95% CI 2-sided [-1.58 to 0.87] — Comparison of iAUC(0-13)
Statistical Analysis 10: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.136, 95% CI 2-sided [-1.41 to 1.13] — Comparison of iAUC(0-13)
Statistical Analysis 11: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.091, 95% CI 2-sided [-1.36 to 1.18] — Comparison of iAUC(0-13)
Statistical Analysis 12: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.206, 95% CI 2-sided [-1.33 to 0.91] — Comparison of iAUC(0-13)
Statistical Analysis 13: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.499, 95% CI 2-sided [-1.68 to 0.68] — Comparison of iAUC(0-24)
Statistical Analysis 14: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-1.24 to 1.21] — Comparison of iAUC(0-24)
Statistical Analysis 15: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.247, 95% CI 2-sided [-1.44 to 0.95] — Comparison of iAUC(0-24)
Statistical Analysis 16: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.661, 95% CI 2-sided [-1.72 to 0.40] — Comparison of iAUC(0-24)

25. Primary Outcome: Part A: Summary of the AUC 0-12 and iAUC 0-12 of Glucagon, Glucagon-like Peptide (GLP; Active and Total)-1, C-peptide, Total Glucose-dependent Insulinotropic Peptide (GIP) and Total Peptide Tyrosine-tyrosine (PYY) and AUC 0-13 and iAUC 0-13 of Insulin
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. For lunch and evening meal in Part A, samples were collected just before the meal and at the following times after starting each meal: 0.5, 1, 1.5 (except breakfast in Part B), 2 and 3 hours. When this results in multiple samples at the same time point, only one sample was collected. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pico moles per Liter
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Pico moles per Liter
  C-peptide, AUC 0-12 | 1533.54 (32.331) | 1518.81 (31.728) | 1523.99 (26.370) | 1513.90 (23.322) | 1418.12 (31.849)
  C-peptide, iAUC 0-12 | 920.62 (34.611) | 874.41 (39.842) | 821.46 (34.785) | 846.34 (29.692) | 836.98 (35.373)
  GIP total, AUC 0-12 | 39.99 (23.579) | 44.91 (28.596) | 44.07 (26.903) | 51.21 (26.338) | 32.76 (28.341)
  GIP total, iAUC 0-12 | 35.36 (25.387) | 38.77 (29.579) | 38.52 (28.757) | 42.15 (24.080) | 28.03 (31.909)
  GLP-1 active, AUC 0-12: number analyzed (Participants) | 10 | 12 | 12 | 11 | 13
  GLP-1 active, AUC 0-12 | 2.14 (1.291) | 2.12 (0.815) | 2.26 (10.182) | 2.20 (7.629) | 5.35 (30.858)
  GLP-1 active, iAUC 0-12: number analyzed (Participants) | 10 | 12 | 12 | 11 | 13
  GLP-1 active, iAUC 0-12 | 0.05 (172.301) | 0.06 (346.410) | 0.12 (153.295) | 0.07 (191.029) | 3.05 (50.439)
  GLP-1 total, AUC 0-12 | 5.66 (34.886) | 5.83 (41.037) | 6.13 (29.049) | 7.44 (39.162) | 4.04 (39.915)
  GLP-1 total, iAUC 0-12 | 3.35 (54.162) | 3.34 (57.021) | 3.64 (42.846) | 4.33 (41.068) | 2.36 (71.247)
  Glucagon, AUC 0-12: number analyzed (Participants) | 6 | 7 | 8 | 9 | 8
  Glucagon, AUC 0-12 | 8.11 (27.492) | 9.55 (39.783) | 10.62 (37.541) | 9.34 (52.831) | 7.44 (37.297)
  Glucagon, iAUC 0-12: number analyzed (Participants) | 6 | 7 | 8 | 9 | 8
  Glucagon, iAUC 0-12 | 3.77 (54.721) | 2.81 (194.661) | 2.60 (148.080) | 1.97 (83.805) | 1.86 (50.802)
  Insulin, AUC 0-13 | 267.68 (63.475) | 272.04 (45.425) | 277.10 (53.966) | 280.90 (46.494) | 210.66 (48.374)
  Insulin, iAUC 0-13 | 211.95 (64.157) | 199.42 (46.245) | 207.02 (55.393) | 208.19 (50.315) | 151.53 (51.789)
  PYY total, AUC 0-12 | 23.04 (30.099) | 29.72 (26.567) | 30.46 (34.393) | 35.38 (34.413) | 17.67 (32.393)
  PYY total, iAUC 0-12 | 10.34 (45.444) | 15.04 (38.723) | 15.56 (54.028) | 17.74 (43.836) | 3.79 (105.916)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -49.898, 95% CI 2-sided [-479.74 to 379.94] — Comparison of C-peptide, AUC 0-12
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -61.642, 95% CI 2-sided [-507.32 to 384.04] — Comparison of C-peptide, AUC 0-12
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -85.849, 95% CI 2-sided [-530.07 to 358.37] — Comparison of C-peptide, AUC 0-12
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -101.422, 95% CI 2-sided [-494.09 to 291.25] — Comparison of C-peptide, AUC 0-12
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -39.239, 95% CI 2-sided [-340.32 to 261.85] — Comparison of C-peptide, iAUC 0-12
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -117.435, 95% CI 2-sided [-429.61 to 194.74] — Comparison of C-peptide, iAUC 0-12
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -121.982, 95% CI 2-sided [-433.14 to 189.18] — Comparison of C-peptide, iAUC 0-12
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -81.016, 95% CI 2-sided [-356.07 to 194.03] — Comparison of C-peptide, iAUC 0-12
Statistical Analysis 9: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.812, 95% CI 2-sided [-8.08 to 13.70] — Comparison of GIP total, AUC 0-12
Statistical Analysis 10: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.023, 95% CI 2-sided [-8.27 to 14.32] — Comparison of GIP total, AUC 0-12
Statistical Analysis 11: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 11.483, 95% CI 2-sided [0.23 to 22.74] — Comparison of GIP total, AUC 0-12
Statistical Analysis 12: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -7.093, 95% CI 2-sided [-17.04 to 2.86] — Comparison of GIP total, AUC 0-12
Statistical Analysis 13: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.500, 95% CI 2-sided [-7.28 to 12.28] — Comparison of GIP total, iAUC 0-12
Statistical Analysis 14: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.526, 95% CI 2-sided [-6.61 to 13.67] — Comparison of GIP total, iAUC 0-12
Statistical Analysis 15: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.934, 95% CI 2-sided [-2.17 to 18.04] — Comparison of GIP total, iAUC 0-12
Statistical Analysis 16: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -7.055, 95% CI 2-sided [-15.99 to 1.88] — Comparison of GIP total, iAUC 0-12
Statistical Analysis 17: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.79 to 0.76] — Comparison of GLP-1 active, AUC 0-12
Statistical Analysis 18: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.78 to 0.82] — Comparison of GLP-1 active, AUC 0-12
Statistical Analysis 19: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.78 to 0.85] — Comparison of GLP-1 active, AUC 0-12
Statistical Analysis 20: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.454, 95% CI 2-sided [2.74 to 4.17] — Comparison of GLP-1 active, AUC 0-12
Statistical Analysis 21: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.78 to 0.75] — Comparison of GLP-1 active, iAUC 0-12
Statistical Analysis 22: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.79 to 0.80] — Comparison of GLP-1 active, iAUC 0-12
Statistical Analysis 23: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.79 to 0.83] — Comparison of GLP-1 active, iAUC 0-12
Statistical Analysis 24: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.399, 95% CI 2-sided [2.69 to 4.11] — Comparison of GLP-1 active, iAUC 0-12
Statistical Analysis 25: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-2.06 to 2.17] — Comparison of GLP-1 total, AUC 0-12
Statistical Analysis 26: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.223, 95% CI 2-sided [-1.97 to 2.42] — Comparison of GLP-1 total, AUC 0-12
Statistical Analysis 27: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.835, 95% CI 2-sided [-0.35 to 4.02] — Comparison of GLP-1 total, AUC 0-12
Statistical Analysis 28: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.629, 95% CI 2-sided [-3.56 to 0.30] — Comparison of GLP-1 total, AUC 0-12
Statistical Analysis 29: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [-1.70 to 1.86] — Comparison of GLP-1 total, iAUC 0-12
Statistical Analysis 30: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.286, 95% CI 2-sided [-1.56 to 2.13] — Comparison of GLP-1 total, iAUC 0-12
Statistical Analysis 31: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.764, 95% CI 2-sided [-1.08 to 2.60] — Comparison of GLP-1 total, iAUC 0-12
Statistical Analysis 32: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.336, 95% CI 2-sided [-2.96 to 0.29] — Comparison of GLP-1 total, iAUC 0-12
Statistical Analysis 33: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority; Mean Difference (Final Values) = 0.962, 95% CI 2-sided [-4.26 to 6.18] — Comparison of Glucagon, AUC 0-12
Statistical Analysis 34: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.067, 95% CI 2-sided [-2.56 to 8.69] — Comparison of Glucagon, AUC 0-12
Statistical Analysis 35: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.517, 95% CI 2-sided [-2.98 to 8.01] — Comparison of Glucagon, AUC 0-12
Statistical Analysis 36: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.714, 95% CI 2-sided [-5.56 to 4.13] — Comparison of Glucagon, AUC 0-12
Statistical Analysis 37: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.866, 95% CI 2-sided [-6.40 to 0.67] — Comparison of Glucagon, iAUC 0-12
Statistical Analysis 38: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.865, 95% CI 2-sided [-4.68 to 2.95] — Comparison of Glucagon, iAUC 0-12
Statistical Analysis 39: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.436, 95% CI 2-sided [-4.16 to 3.29] — Comparison of Glucagon, iAUC 0-12
Statistical Analysis 40: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.573, 95% CI 2-sided [-4.86 to 1.71] — Comparison of Glucagon, iAUC 0-12
Statistical Analysis 41: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -24.740, 95% CI 2-sided [-168.38 to 118.90] — Comparison of Insulin, AUC 0-13
Statistical Analysis 42: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -12.229, 95% CI 2-sided [-161.16 to 136.70] — Comparison of Insulin, AUC 0-13
Statistical Analysis 43: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -9.628, 95% CI 2-sided [-158.07 to 138.81] — Comparison of Insulin, AUC 0-13
Statistical Analysis 44: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -66.936, 95% CI 2-sided [-198.15 to 64.28] — Comparison of Insulin, AUC 0-13
Statistical Analysis 45: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -36.042, 95% CI 2-sided [-150.57 to 78.48] — Comparison of Insulin, iAUC 0-13
Statistical Analysis 46: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -22.525, 95% CI 2-sided [-141.27 to 96.22] — Comparison of Insulin, iAUC 0-13
Statistical Analysis 47: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -22.000, 95% CI 2-sided [-140.36 to 96.36] — Comparison of Insulin, iAUC 0-13
Statistical Analysis 48: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -66.324, 95% CI 2-sided [-170.95 to 38.30] — Comparison of Insulin, iAUC 0-13
Statistical Analysis 49: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 5.982, 95% CI 2-sided [-2.66 to 14.62] — Comparison of PYY total, AUC 0-12
Statistical Analysis 50: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 8.908, 95% CI 2-sided [-0.05 to 17.86] — Comparison of PYY total, AUC 0-12
Statistical Analysis 51: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 14.317, 95% CI 2-sided [5.39 to 23.24] — Comparison of PYY total, AUC 0-12
Statistical Analysis 52: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -5.440, 95% CI 2-sided [-13.33 to 2.45] — Comparison of PYY total, AUC 0-12
Statistical Analysis 53: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 4.999, 95% CI 2-sided [-1.87 to 11.87] — Comparison of PYY total, iAUC 0-12
Statistical Analysis 54: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.909, 95% CI 2-sided [-0.22 to 14.03] — Comparison of PYY total, iAUC 0-12
Statistical Analysis 55: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 9.036, 95% CI 2-sided [1.93 to 16.14] — Comparison of PYY total, iAUC 0-12
Statistical Analysis 56: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -6.390, 95% CI 2-sided [-12.67 to -0.11] — Comparison of PYY total, iAUC 0-12

26. Primary Outcome: Part A: Summary of the OGTT AUC (0-3) and iAUC(0-3)-Glucose
Description: Blood samples for the determination of glucose were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. When this results in multiple samples at the same time point, only one sample was collected. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millimoles per Liter
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Millimoles per Liter
  AUC 0-3 | 12.82 (14.080) | 12.79 (18.904) | 12.12 (16.572) | 11.26 (16.651) | 11.97 (25.950)
  iAUC 0-3 | 5.55 (16.251) | 5.17 (19.811) | 4.78 (20.419) | 4.25 (27.727) | 4.43 (28.677)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.564, 95% CI 2-sided [-2.69 to 1.56] — Comparison of AUC 0-3
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.846, 95% CI 2-sided [-3.05 to 1.36] — Comparison of AUC 0-3
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.175, 95% CI 2-sided [-3.37 to 1.02] — Comparison of AUC 0-3
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.617, 95% CI 2-sided [-2.56 to 1.33] — Comparison of AUC 0-3
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.626, 95% CI 2-sided [-1.64 to 0.39] — Comparison of iAUC 0-3
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.956, 95% CI 2-sided [-2.01 to 0.09] — Comparison of iAUC 0-3
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.103, 95% CI 2-sided [-2.15 to -0.06] — Comparison of iAUC 0-3
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.990, 95% CI 2-sided [-1.91 to -0.07] — Comparison of iAUC 0-3

27. Primary Outcome: Part A: Summary of the OGTT AUC (0-2) and iAUC(0-2)- C-peptide, Total GIP, GLP-1 (Active and Total), Glucagon and Total PYY and AUC 0-3 and iAUC 0-3 of Insulin
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. When this results in multiple samples at the same time point, only one sample was collected. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pico moles per Liter
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Pico moles per Liter
  C-peptide, AUC 0-2 | 1207.17 (27.472) | 1352.32 (28.098) | 1357.81 (20.421) | 1387.78 (25.473) | 1287.66 (34.527)
  C-peptide, iAUC 0-2 | 563.75 (46.497) | 676.24 (40.442) | 620.95 (41.762) | 695.31 (43.060) | 692.11 (45.456)
  GIP total, AUC 0-2 | 29.73 (34.698) | 37.86 (26.719) | 34.82 (34.834) | 42.25 (34.507) | 26.57 (40.429)
  GIP total, iAUC 0-2 | 25.30 (36.096) | 31.50 (30.146) | 29.27 (37.728) | 33.51 (29.808) | 21.79 (45.161)
  GLP-1 active, AUC 0-2 | 2.12 (0.426) | 2.12 (0.000) | 2.18 (4.606) | 2.14 (2.540) | 4.73 (22.230)
  GLP-1 active, iAUC 0-2 | 0.03 (331.662) | NA (NA) — NA indicates data not evaluable. | 0.18 (158.801) | 0.18 (331.662) | 2.47 (38.584)
  GLP-1 total, AUC 0-2 | 4.45 (32.218) | 4.51 (36.731) | 5.02 (27.985) | 5.59 (37.459) | 2.97 (34.891)
  GLP-1 total, iAUC 0-2 | 2.65 (49.892) | 1.66 (80.669) | 2.40 (51.939) | 2.38 (49.604) | 1.26 (63.785)
  Glucagon, AUC 0-2: number analyzed (Participants) | 7 | 11 | 11 | 7 | 9
  Glucagon, AUC 0-2 | 3.60 (41.288) | 4.77 (40.537) | 6.08 (39.006) | 4.49 (44.216) | 3.85 (62.260)
  Glucagon, iAUC 0-2: number analyzed (Participants) | 7 | 11 | 11 | 7 | 9
  Glucagon, iAUC 0-2 | 0.56 (448.254) | 0.24 (-157.518) | 0.62 (-157.616) | 0.73 (-122.368) | 0.39 (-121.494)
  Insulin, AUC 0-3 | 204.77 (46.353) | 230.91 (39.743) | 235.88 (42.743) | 254.61 (50.810) | 213.17 (49.480)
  Insulin, iAUC 0-3 | 146.03 (52.193) | 156.32 (41.131) | 161.05 (45.743) | 179.93 (58.350) | 150.33 (56.399)
  PYY total, AUC 0-2 | 16.76 (23.007) | 19.30 (42.059) | 22.45 (39.164) | 23.42 (25.206) | 13.93 (35.971)
  PYY total, iAUC 0-2 | 5.89 (62.399) | 4.66 (95.556) | 6.81 (74.605) | 5.59 (62.823) | 1.25 (162.044)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 152.962, 95% CI 2-sided [-200.57 to 506.49] — Comparison of C-peptide, AUC 0-2
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 113.866, 95% CI 2-sided [-252.69 to 480.42] — Comparison of C-peptide, AUC 0-2
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 114.474, 95% CI 2-sided [-250.89 to 479.83] — Comparison of C-peptide, AUC 0-2
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 136.638, 95% CI 2-sided [-186.32 to 459.60] — Comparison of C-peptide, AUC 0-2
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 163.622, 95% CI 2-sided [-127.31 to 454.55] — Comparison of C-peptide, iAUC 0-2
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 58.074, 95% CI 2-sided [-243.57 to 359.72] — Comparison of C-peptide, iAUC 0-2
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 78.341, 95% CI 2-sided [-222.32 to 379.00] — Comparison of C-peptide, iAUC 0-2
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 157.044, 95% CI 2-sided [-108.73 to 422.82] — Comparison of C-peptide, iAUC 0-2
Statistical Analysis 9: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.539, 95% CI 2-sided [-4.79 to 17.87] — Comparison of GIP total, AUC 0-2
Statistical Analysis 10: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 4.095, 95% CI 2-sided [-7.65 to 15.84] — Comparison of GIP total, AUC 0-2
Statistical Analysis 11: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 13.033, 95% CI 2-sided [1.33 to 24.74] — Comparison of GIP total, AUC 0-2
Statistical Analysis 12: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.824, 95% CI 2-sided [-13.17 to 7.52] — Comparison of GIP total, AUC 0-2
Statistical Analysis 13: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.227, 95% CI 2-sided [-3.47 to 15.93] — Comparison of GIP total, iAUC 0-2
Statistical Analysis 14: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 4.598, 95% CI 2-sided [-5.46 to 14.65] — Comparison of GIP total, iAUC 0-2
Statistical Analysis 15: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 9.484, 95% CI 2-sided [-0.54 to 19.51] — Comparison of GIP total, iAUC 0-2
Statistical Analysis 16: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.786, 95% CI 2-sided [-11.65 to 6.08] — Comparison of GIP total, iAUC 0-2
Statistical Analysis 17: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [-0.38 to 0.52] — Comparison of GLP-1 active, AUC 0-2
Statistical Analysis 18: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.256, 95% CI 2-sided [-0.21 to 0.72] — Comparison of GLP-1 active, AUC 0-2
Statistical Analysis 19: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.42 to 0.51] — Comparison of GLP-1 active, AUC 0-2
Statistical Analysis 20: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.694, 95% CI 2-sided [2.28 to 3.11] — Comparison of GLP-1 active, AUC 0-2
Statistical Analysis 21: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.36 to 0.50] — Comparison of GLP-1 active, iAUC 0-2
Statistical Analysis 22: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.243, 95% CI 2-sided [-0.20 to 0.69] — Comparison of GLP-1 active, iAUC 0-2
Statistical Analysis 23: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.41 to 0.47] — Comparison of GLP-1 active, iAUC 0-2
Statistical Analysis 24: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.643, 95% CI 2-sided [2.25 to 3.04] — Comparison of GLP-1 active, iAUC 0-2
Statistical Analysis 25: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.055, 95% CI 2-sided [-1.44 to 1.55] — Comparison of GLP-1 total, AUC 0-2
Statistical Analysis 26: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.268, 95% CI 2-sided [-1.28 to 1.82] — Comparison of GLP-1 total, AUC 0-2
Statistical Analysis 27: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.894, 95% CI 2-sided [-0.65 to 2.44] — Comparison of GLP-1 total, AUC 0-2
Statistical Analysis 28: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.483, 95% CI 2-sided [-2.85 to -0.12] — Comparison of GLP-1 total, AUC 0-2
Statistical Analysis 29: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.081, 95% CI 2-sided [-1.18 to 1.34] — Comparison of GLP-1 total, iAUC 0-2
Statistical Analysis 30: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.331, 95% CI 2-sided [-0.97 to 1.63] — Comparison of GLP-1 total, iAUC 0-2
Statistical Analysis 31: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.177, 95% CI 2-sided [-1.48 to 1.12] — Comparison of GLP-1 total, iAUC 0-2
Statistical Analysis 32: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Median Difference (Final Values) = -1.190, 95% CI 2-sided [-2.34 to -0.04] — Comparison of GLP-1 total, iAUC 0-2
Statistical Analysis 33: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.235, 95% CI 2-sided [-1.51 to 3.98] — Comparison of Glucagon, AUC 0-2
Statistical Analysis 34: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.877, 95% CI 2-sided [0.04 to 5.71] — Comparison of Glucagon, AUC 0-2
Statistical Analysis 35: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.473, 95% CI 2-sided [-1.21 to 4.16] — Comparison of Glucagon, AUC 0-2
Statistical Analysis 36: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.274, 95% CI 2-sided [-2.20 to 2.74] — Comparison of Glucagon, AUC 0-2
Statistical Analysis 37: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.177, 95% CI 2-sided [-4.92 to 0.56] — Comparison of Glucagon, iAUC 0-2
Statistical Analysis 38: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.909, 95% CI 2-sided [-4.74 to 0.93] — Comparison of Glucagon, iAUC 0-2
Statistical Analysis 39: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.053, 95% CI 2-sided [-3.74 to 1.63] — Comparison of Glucagon, iAUC 0-2
Statistical Analysis 40: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.249, 95% CI 2-sided [-3.72 to 1.22] — Comparison of Glucagon, iAUC 0-2
Statistical Analysis 41: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 13.389, 95% CI 2-sided [-95.82 to 122.59] — Comparison of Insulin, AUC 0-3
Statistical Analysis 42: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 9.980, 95% CI 2-sided [-103.25 to 123.21] — Comparison of Insulin, AUC 0-3
Statistical Analysis 43: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 32.426, 95% CI 2-sided [-80.43 to 145.28] — Comparison of Insulin, AUC 0-3
Statistical Analysis 44: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 22.994, 95% CI 2-sided [-76.77 to 122.76] — Comparison of Insulin, AUC 0-3
Statistical Analysis 45: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.088, 95% CI 2-sided [-86.79 to 90.97] — Comparison of Insulin, iAUC 0-3
Statistical Analysis 46: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.316, 95% CI 2-sided [-92.47 to 91.84] — Comparison of Insulin, iAUC 0-3
Statistical Analysis 47: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 20.053, 95% CI 2-sided [-71.80 to 111.91] — Comparison of Insulin, iAUC 0-3
Statistical Analysis 48: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 23.606, 95% CI 2-sided [-57.59 to 104.80] — Comparison of Insulin, iAUC 0-3
Statistical Analysis 49: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.506, 95% CI 2-sided [-3.13 to 10.14] — Comparison of PYY total, AUC 0-2
Statistical Analysis 50: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.295, 95% CI 2-sided [0.41 to 14.18] — Comparison of PYY total, AUC 0-2
Statistical Analysis 51: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.006, 95% CI 2-sided [0.15 to 13.87] — Comparison of PYY total, AUC 0-2
Statistical Analysis 52: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.555, 95% CI 2-sided [-8.62 to 3.51] — Comparison of PYY total, AUC 0-2
Statistical Analysis 53: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.523, 95% CI 2-sided [-2.13 to 7.17] — Comparison of PYY total, iAUC 0-2
Statistical Analysis 54: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 5.296, 95% CI 2-sided [0.47 to 10.12] — Comparison of PYY total, iAUC 0-2
Statistical Analysis 55: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.726, 95% CI 2-sided [-3.08 to 6.53] — Comparison of PYY total, iAUC 0-2
Statistical Analysis 56: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -3.506, 95% CI 2-sided [-7.75 to 0.74] — Comparison of PYY total, iAUC 0-2

28. Primary Outcome: Part A: Summary of the OGTT Derived Parameters: Disposition Index
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. When this results in multiple samples at the same time point, only one sample was collected. It was calculated by multiplying insulin glucose index with insulin sensitivity index. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [(µIU/mL)/(mg/deciliter [dL])]^2
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
[(µIU/mL)/(mg/deciliter [dL])]^2 | 0.87 (201.883) | 0.76 (65.975) | 1.07 (78.991) | 0.94 (62.371) | 0.86 (95.526)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.241, 95% CI 2-sided [-0.84 to 1.32]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.523, 95% CI 2-sided [-0.60 to 1.64]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.053, 95% CI 2-sided [-1.17 to 1.06]
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [-0.81 to 1.16]

29. Primary Outcome: Part A: Summary of the OGTT Derived Parameters: Glucose/Insulin and Insulin/Glucose Ratio
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. When this results in multiple samples at the same time point, only one sample was collected. It was calculated as insulin/glucose ratio was calculated as insulin AUC(0-3]/glucose AUC(0-3) during OGTT, while glucose/insulin ratio was calculated as glucose AUC(0-3)/insulin AUC(0-3) during OGTT. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
Ratio
  G/I ratio | 0.06 (60.128) | 0.06 (73.172) | 0.05 (61.602) | 0.04 (56.203) | 0.06 (154.204)
  I/G ratio | 15.98 (47.582) | 18.05 (40.272) | 19.46 (50.494) | 22.61 (60.152) | 17.80 (54.449)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.010, 95% CI 2-sided [-0.08 to 0.06] — Comparison of G/I ratio
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.07 to 0.07] — Comparison of G/I ratio
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.07 to 0.07] — Comparison of G/I ratio
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.04 to 0.08] — Comparison of G/I ratio
Statistical Analysis 5: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.269, 95% CI 2-sided [-8.31 to 12.85] — Comparison of I/G ratio
Statistical Analysis 6: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.959, 95% CI 2-sided [-8.01 to 13.93] — Comparison of I/G ratio
Statistical Analysis 7: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.053, 95% CI 2-sided [-4.88 to 16.99] — Comparison of I/G ratio
Statistical Analysis 8: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 4.017, 95% CI 2-sided [-5.65 to 13.68] — Comparison of I/G ratio

30. Primary Outcome: Part A: Summary of the OGTT Derived Parameters: Insulin Glucose Index
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. When this results in multiple samples at the same time point, only one sample was collected. It was calculated as insulin (30 min) - insulin (0 min)/glucose (30 min) - glucose (0 min). It was calculated as insulin (30 min) - insulin (0 min)/glucose (30 min) - glucose (0 min). The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µIU/mL/mg/dL
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
µIU/mL/mg/dL | 0.23 (144.722) | 0.22 (54.340) | 0.28 (67.645) | 0.26 (64.622) | 0.21 (75.325)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.025, 95% CI 2-sided [-0.28 to 0.22] — Comparison of insulin glucose index
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.055, 95% CI 2-sided [-0.20 to 0.31] — Comparison of insulin glucose index
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.29 to 0.23] — Comparison of insulin glucose index
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.041, 95% CI 2-sided [-0.27 to 0.19] — Comparison of insulin glucose index

31. Primary Outcome: Part A: Summary of the OGTT Derived Parameters: Insulin Sensitivity Index
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. When this results in multiple samples at the same time point, only one sample was collected. It was calculated as 10,000/square root ([mean plasma insulin × mean plasma glucose during OGTT or meal challenge] × [fasting plasma glucose × fasting plasma insulin]). The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Up to Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/(mg/dL)×1/(µIU/mL)
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg | Part A: GSK1292263 150 mg | Part A: GSK1292263 800 mg | Part A: Sitagliptin 100 mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 13
1/(mg/dL)×1/(µIU/mL) | 3.95 (44.078) | 3.47 (45.993) | 3.87 (42.720) | 3.60 (37.292) | 4.01 (47.046)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: GSK1292263 25 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.346, 95% CI 2-sided [-2.06 to 1.37]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: GSK1292263 150 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-1.82 to 1.73]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: GSK1292263 800 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.388, 95% CI 2-sided [-2.16 to 1.38]
Statistical Analysis 4: Comparison: Part A: Placebo vs Part A: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.133, 95% CI 2-sided [-1.43 to 1.70]

32. Primary Outcome: Part C: Summary of Change From Baseline in Fasted Glucose
Description: Blood samples were collected fasting pre-breakfast and pre-morning dose (PD time 0) on Days -1, 13 and 14 and then at 10, 20, 30, 60, 90, 120, 180 min after eating the standardized breakfast meal tolerance test. For lunch (4 hour post-morning dose) samples were collected just before the meal and after starting each meal: 0.5, 1, 1.5, 2 and 3 hours. For the evening meal (10 hour post-morning dose), BID dosing groups followed the sequence of sampling, food and dosing as for breakfast (PD sample immediately before meal, eat and then dose), then 0.5, 1, 1.5, 2 and 3 hours post-dinner. A sample was also collected 24 hours post-dose. When this results in multiple samples at the same time point, only one sample was collected. Change from Baseline was calculated by subtracting Baseline value minus post-Baseline value. The point estimates and corresponding 95% CI for treatment ratios were calculated for treatment comparisons versus placebo.
Time Frame: Baseline (Day 1 pre-dose) and Day -1, 13 and 14.
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millimoles per Liter
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 12
Millimoles per Liter
  Day 7, 1 Hour | 4.60 (73.478) | 4.93 (41.905) | 7.39 (36.730) | 5.17 (57.754) | 5.51 (38.497) | 4.09 (70.342)
  Day 7, 2 Hours | 4.71 (150.720) | 3.65 (82.667) | 5.00 (45.953) | 3.61 (75.258) | 2.59 (60.658) | 3.17 (152.623)
  Day 7, 4 Hours | 1.85 (-482.690) | 1.11 (-606.064) | 1.13 (270.863) | 2.05 (685.731) | 0.95 (-223.367) | 2.13 (-188.101)
  Day 7, 6 Hours | 4.98 (75.579) | 3.72 (67.064) | 6.16 (51.414) | 4.15 (74.614) | 3.93 (62.647) | 3.70 (270.326)
  Day 7, 10 Hours | 2.07 (271.597) | 1.91 (166.934) | 3.18 (83.271) | 3.13 (133.236) | 2.06 (228.901) | 5.17 (-1115.737)
  Day 7, 12 Hours | 3.66 (105.362) | 2.42 (71.838) | 4.41 (49.106) | 3.53 (82.377) | 3.77 (60.670) | 3.33 (119.827)
  Day 14, 24 Hours | 1.26 (-1044.892) | 1.09 (3884.234) | 1.34 (179.562) | 1.21 (2819.220) | 1.52 (565.287) | 2.08 (-323.555)
Statistical Analysis 1: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.523, 95% CI 2-sided [-3.04 to 2.00] — Comparison of Day 7, 1 Hour
Statistical Analysis 2: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.569, 95% CI 2-sided [-3.07 to 1.94] — Comparison of Day 7, 1 Hour
Statistical Analysis 3: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 2.064, 95% CI 2-sided [-0.45 to 4.57] — Comparison of Day 7, 1 Hour
Statistical Analysis 4: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.316, 95% CI 2-sided [-2.19 to 2.82] — Comparison of Day 7, 1 Hour
Statistical Analysis 5: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -1.484, 95% CI 2-sided [-3.99 to 1.02] — Comparison of Day 7, 1 Hour
Statistical Analysis 6: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.795, 95% CI 2-sided [-3.27 to 1.68] — Comparison of Day 7, 2 Hours
Statistical Analysis 7: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.313, 95% CI 2-sided [-2.78 to 2.15] — Comparison of Day 7, 2 Hours
Statistical Analysis 8: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 2.441, 95% CI 2-sided [-0.03 to 4.91] — Comparison of Day 7, 2 Hours
Statistical Analysis 9: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.884, 95% CI 2-sided [-1.58 to 3.34] — Comparison of Day 7, 2 Hours
Statistical Analysis 10: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -1.222, 95% CI 2-sided [-3.69 to 1.24] — Comparison of Day 7, 2 Hours
Statistical Analysis 11: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.017, 95% CI 2-sided [-2.06 to 2.03] — Comparison of Day 7, 4 Hours
Statistical Analysis 12: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.475, 95% CI 2-sided [-1.56 to 2.51] — Comparison of Day 7, 4 Hours
Statistical Analysis 13: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 1.512, 95% CI 2-sided [-0.53 to 3.55] — Comparison of Day 7, 4 Hours
Statistical Analysis 14: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 1.233, 95% CI 2-sided [-0.80 to 3.26] — Comparison of Day 7, 4 Hours
Statistical Analysis 15: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -1.011, 95% CI 2-sided [-3.05 to 1.02] — Comparison of Day 7, 4 Hours
Statistical Analysis 16: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.189, 95% CI 2-sided [-3.05 to 2.67] — Comparison of Day 7, 6 Hours
Statistical Analysis 17: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.456, 95% CI 2-sided [-2.39 to 3.30] — Comparison of Day 7, 6 Hours
Statistical Analysis 18: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 2.706, 95% CI 2-sided [-0.14 to 5.56] — Comparison of Day 7, 6 Hours
Statistical Analysis 19: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 1.062, 95% CI 2-sided [-1.78 to 3.91] — Comparison of Day 7, 6 Hours
Statistical Analysis 20: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -2.708, 95% CI 2-sided [-5.55 to 0.14] — Comparison of Day 7, 6 Hours
Statistical Analysis 21: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.147, 95% CI 2-sided [-2.41 to 2.70] — Comparison of Day 7, 10 Hours
Statistical Analysis 22: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.452, 95% CI 2-sided [-2.09 to 2.99] — Comparison of Day 7, 10 Hours
Statistical Analysis 23: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 2.418, 95% CI 2-sided [-0.13 to 4.96] — Comparison of Day 7, 10 Hours
Statistical Analysis 24: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 1.063, 95% CI 2-sided [-1.47 to 3.60] — Comparison of Day 7, 10 Hours
Statistical Analysis 25: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -1.509, 95% CI 2-sided [-4.05 to 1.03] — Comparison of Day 7, 10 Hours
Statistical Analysis 26: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -1.300, 95% CI 2-sided [-4.20 to 1.60] — Comparison of Day 7, 12 Hours
Statistical Analysis 27: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -1.325, 95% CI 2-sided [-4.21 to 1.56] — Comparison of Day 7, 12 Hours
Statistical Analysis 28: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 1.000, 95% CI 2-sided [-1.89 to 3.89] — Comparison of Day 7, 12 Hours
Statistical Analysis 29: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.265, 95% CI 2-sided [-3.14 to 2.62] — Comparison of Day 7, 12 Hours
Statistical Analysis 30: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.516, 95% CI 2-sided [-3.40 to 2.37] — Comparison of Day 7, 12 Hours
Statistical Analysis 31: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.515, 95% CI 2-sided [-2.29 to 1.26] — Comparison of Day 14, 24 Hours
Statistical Analysis 32: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.225, 95% CI 2-sided [-1.99 to 1.55] — Comparison of Day 14, 24 Hours
Statistical Analysis 33: Comparison: Part C: GSK1292263 300 mg BID; Test type: Superiority or Other; Mean Difference (Net) = 0.501, 95% CI 2-sided [-1.28 to 2.28] — Comparison of Day 14, 24 Hours
Statistical Analysis 34: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.168, 95% CI 2-sided [-1.98 to 1.65] — Comparison of Day 14, 24 Hours
Statistical Analysis 35: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -1.043, 95% CI 2-sided [-2.81 to 0.73] — Comparison of Day 14, 24 Hours

33. Primary Outcome: Part C: Summary of Change From Baseline in Fasted Insulin
Description: as for outcome 32
Time Frame: Baseline (Day 1 pre-dose) and Day -1, 13 and 14
Population: The PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millimoles per Liter
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 12
Millimoles per Liter
  Day 7, 1 Hour | 158.91 (115.808) | 117.15 (53.056) | 151.56 (88.163) | 129.44 (101.186) | 216.95 (91.593) | 162.83 (62.028)
  Day 7, 2 Hours | 92.17 (99.479) | 94.18 (55.907) | 143.75 (108.953) | 87.30 (145.016) | 160.57 (123.482) | 163.46 (80.530)
  Day 7, 4 Hours | 35.05 (650.532) | 20.10 (354.147) | 27.32 (97.622) | 21.93 (337.965) | 19.41 (150.506) | 30.25 (169.388)
  Day 7, 6 Hours | 103.52 (76.383) | 88.70 (70.484) | 136.15 (92.906) | 131.08 (84.834) | 142.10 (74.418) | 130.88 (48.541)
  Day 7, 10 Hours | 68.08 (129.341) | 55.28 (131.603) | 55.40 (86.768) | 66.90 (162.220) | 64.04 (72.943) | 39.35 (76.204)
  Day 7, 12 Hours | 107.52 (77.742) | 95.16 (69.323) | 98.26 (140.843) | 114.93 (81.742) | 138.42 (54.450) | 123.65 (74.446)
  Day 14, 24 Hours | 12.45 (-180.869) | 1.51 (-256.494) | 3.54 (-116.769) | 11.03 (-226.913) | 7.87 (-322.274) | 3.26 (-191.100)
Statistical Analysis 1: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -70.457, 95% CI 2-sided [-214.72 to 73.80] — Day 7, 1 Hour
Statistical Analysis 2: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -151.722, 95% CI 2-sided [-295.98 to -7.46] — Day 7, 1 Hour
Statistical Analysis 3: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -69.113, 95% CI 2-sided [-213.48 to 75.25] — Day 7, 1 Hour
Statistical Analysis 4: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -104.468, 95% CI 2-sided [-248.72 to 39.78] — Day 7, 1 Hour
Statistical Analysis 5: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -118.462, 95% CI 2-sided [-263.93 to 27.01] — Day 7, 1 Hour
Statistical Analysis 6: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -114.340, 95% CI 2-sided [-264.78 to 36.10] — Day 7, 2 Hours
Statistical Analysis 7: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -116.462, 95% CI 2-sided [-266.90 to 33.98] — Day 7, 2 Hours
Statistical Analysis 8: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -4.201, 95% CI 2-sided [-154.75 to 146.35] — Day 7, 2 Hours
Statistical Analysis 9: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -48.270, 95% CI 2-sided [-198.70 to 102.16] — Day 7, 2 Hours
Statistical Analysis 10: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -50.605, 95% CI 2-sided [-202.31 to 101.10] — Day 7, 2 Hours
Statistical Analysis 11: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -7.231, 95% CI 2-sided [-40.84 to 26.38] — Day 7, 4 Hours
Statistical Analysis 12: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -5.025, 95% CI 2-sided [-38.63 to 28.58] — Day 7, 4 Hours
Statistical Analysis 13: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 9.523, 95% CI 2-sided [-24.11 to 43.16] — Day 7, 4 Hours
Statistical Analysis 14: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -2.618, 95% CI 2-sided [-36.22 to 30.99] — Day 7, 4 Hours
Statistical Analysis 15: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = 20.800, 95% CI 2-sided [-13.09 to 54.69] — Day 7, 4 Hours
Statistical Analysis 16: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -58.864, 95% CI 2-sided [-156.11 to 38.38] — Day 7, 6 Hours
Statistical Analysis 17: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -77.900, 95% CI 2-sided [-175.15 to 19.35] — Day 7, 6 Hours
Statistical Analysis 18: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 28.323, 95% CI 2-sided [-69.00 to 125.65] — Day 7, 6 Hours
Statistical Analysis 19: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -24.499, 95% CI 2-sided [-121.74 to 72.74] — Day 7, 6 Hours
Statistical Analysis 20: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -59.755, 95% CI 2-sided [-157.82 to 38.31] — Day 7, 6 Hours
Statistical Analysis 21: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.222, 95% CI 2-sided [-69.85 to 69.40] — Day 7, 10 Hours
Statistical Analysis 22: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.222, 95% CI 2-sided [-77.28 to 61.98] — Day 7, 10 Hours
Statistical Analysis 23: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 7.148, 95% CI 2-sided [-62.55 to 76.85] — Day 7, 10 Hours
Statistical Analysis 24: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 32.734, 95% CI 2-sided [-36.89 to 102.36] — Day 7, 10 Hours
Statistical Analysis 25: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -9.760, 95% CI 2-sided [-81.01 to 61.49] — Day 7, 10 Hours
Statistical Analysis 26: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -19.594, 95% CI 2-sided [-123.36 to 84.18] — Day 7, 12 Hours
Statistical Analysis 27: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -46.924, 95% CI 2-sided [-150.69 to 56.85] — Day 7, 12 Hours
Statistical Analysis 28: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = 24.715, 95% CI 2-sided [-79.16 to 128.59] — Day 7, 12 Hours
Statistical Analysis 29: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -7.966, 95% CI 2-sided [-111.73 to 95.80] — Day 7, 12 Hours
Statistical Analysis 30: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = 3.108, 95% CI 2-sided [-103.08 to 109.29] — Day 7, 12 Hours
Statistical Analysis 31: Comparison: Part C: GSK1292263 50 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -10.114, 95% CI 2-sided [-25.12 to 4.89] — Day 14, 24 Hours
Statistical Analysis 32: Comparison: Part C: GSK1292263 150 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -8.718, 95% CI 2-sided [-23.71 to 6.28] — Day 14, 24 Hours
Statistical Analysis 33: Comparison: Part C: GSK1292263 300 mg BID vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.622, 95% CI 2-sided [-15.63 to 14.38] — Day 14, 24 Hours
Statistical Analysis 34: Comparison: Part C: GSK1292263 600 mg Once Daily vs Part C: Placebo; Test type: Superiority or Other; Mean Difference (Net) = -12.454, 95% CI 2-sided [-27.78 to 2.88] — Day 14, 24 Hours
Statistical Analysis 35: Comparison: Part C: Placebo vs Part C: Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Net) = -8.681, 95% CI 2-sided [-24.02 to 6.66] — Day 14, 24 Hours

34. Secondary Outcome: Part B: Number of Participants With AEs and SAEs
Description: as for outcome 9
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: GSK1292263 800 mg Fasted Condition Orally: In this part (Cohort 2), eligible T2DM participants on mono-therapy or sub-maximal anti-diabetic medications washed off these medications for 1 week and received a single dose of GSK1292263 800 mg orally in fasted condition. Before participants in Part B were dosed, the safety and tolerability of GSK1292263 800 mg administered in the fasted state to 9 participants in Part A was reviewed to ensure that it was safe to proceed. In Part B, study drug was administered 30 min after breakfast and lunch and dinner was approximately 4 and 10 hours after dosing.
- Part B: GSK1292263 800 mg Fed Condition Orally: In this part (Cohort 2), eligible T2DM participants on mono-therapy or sub-maximal anti-diabetic medications washed off these medications for 1 week and received a single dose of GSK1292263 800 mg orally in fed condition. Before participants in Part B were dosed, the safety and tolerability of GSK1292263 800 mg administered in the fasted state to 9 participants in Part A was reviewed to ensure that it was safe to proceed. In Part B, study drug was administered 30 min after breakfast and lunch and dinner was approximately 4 and 10 hours after dosing.
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Participants
  Any AE | 0 | 1
  Any SAE | 0 | 0

35. Secondary Outcome: Part B: Number of Participants With Abnormal Hematology Parameters of PCI
Description: Hematology parameters included platelet count, RBC count, MCV, total neutrophils, WBC absolute, MCH, lymphocytes, MCHC, monocytes, hemoglobin, eosinophils, hematocrit, reticulocytes and basophils. It was assessed on Screening, Day -1, 2 (of each treatment period) and Follow-up (7 to 10 days after final discharge). Only those parameters for which at least one value of PCI was reported are summarized. Null data is not presented.
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

36. Secondary Outcome: Part B: Number of Participants With Abnormal Clinical Chemistry Parameters of PCI
Description: Clinical chemistry parameters included BUN, potassium, AST, total and direct bilirubin, creatinine, chloride, ALT, uric acid, glucose fasting, GGT, albumin, sodium, magnesium, phosphorus inorganic, calcium, total CO2, ALP, triglycerides, total cholesterol, LDL cholesterol, free fatty acid (NEFA), HDL cholesterol and total protein. It was assessed on Screening, Day -1, 2 (of each treatment period) and Follow-up (7 to 10 days after final discharge). Only those parameters (Glucose, High) for which at least one value of PCI was reported are summarized. Null data is not presented.
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Participants | 1 | 1

37. Secondary Outcome: Part B: Number of Participants With Significant ECG Abnormalities
Description: Twelve-lead ECGs was obtained in a supine position at each time point during the study using an ECG machine that automatically measured PR, QRS, QT and QTc intervals (QTcB and QTcF). Participants with abnormal clinically significant ECG findings is presented. It was assessed on Screening, Day 1 at pre-dose, 1, 2, 3, 4, 6, 10, 16, 24 hours and Follow-up (7 -10 days after final discharge).
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

38. Secondary Outcome: Part B: Number of Participants With Abnormal Vital Signs of PCI
Description: SBP, DBP and pulse rate measurements were recorded at each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 min. Participants with abnormal clinically significant vital signs findings is presented. It was assessed on Screening, Day -1, 1, 2 (pre-dose, 1, 3, 4, 6, 10, 16 and 24 hours of each treatment period) and Follow-up (7 -10 days after final discharge).
Time Frame: Up to Week 7
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

39. Secondary Outcome: Part B: Summary of Plasma Cmax
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. Blood samples for the determination of PK was collected at on Day 1 of each period: immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13 and 24 hours.
Time Frame: Pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13 and 24 hours on Day 1 of each treatment period.
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per mL
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Nanograms per mL | 339.52 (32.581) | 944.21 (47.330)

40. Secondary Outcome: Part B: Summary of T-max and T-lag
Description: The time at which Cmax was observed was determined directly from the raw concentration-time data. The lag time before observation of drug concentrations in sample matrix determined as the time of the sample preceding the first quantifiable concentration. Blood samples for the determination of PK was collected at on Day 1 of each period: immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13 and 24 hours.
Time Frame: Pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13 and 24 hours on Day 1 of each treatment period
Population: PK Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Hour
  T-max | 2.00 [2.0 to 4.0] | 4.98 [4.0 to 13.1]
  T-lag | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.0]

41. Secondary Outcome: Part B: Summary of AUC0-t and AUC0-24
Description: The AUC 0-24 and AUC 0-t determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples for the determination of PK was collected at on Day 1 of each period: immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13 and 24 hours.
Time Frame: Pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13 and 24 hours on Day 1 of each treatment period
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms×hour per mL
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Nanograms×hour per mL
  AUC 0-24 | 3370.43 (21.507) | 12639.84 (27.622)
  AUC 0-t | 3370.43 (21.507) | 12659.88 (27.391)

42. Secondary Outcome: Part B: Summary of Change From Baseline in Fasted Glucose
Description: Blood samples for the determination of glucose were collected at pre-dose on Day 1 of each dosing period and immediately prior to and at 10, 20, 30, 60, 90, 120, 180 min after administration of the 75 grams glucose drink. For lunch and evening meal in Part A, samples were collected just before the meal and at the following times after starting each meal: 0.5, 1, 1.5 (except breakfast in Part B), 2 and 3 hours. When this results in multiple samples at the same time point, only one sample was collected. Change from Baseline was calculated by subtracting Baseline value from post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 1 (24 hours)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millimoles per Liter
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Millimoles per Liter | 0.40 (62.025) | 1.95 (-10966.01)

43. Secondary Outcome: Part B: Summary of Change From Baseline in Fasted Glucagon, GLP-1, C-peptide, Total GIP, Total PYY and Insulin
Description: Blood samples for the determination of glucose and other PD markers were collected at pre-dose on Day 1 of each dosing period. For breakfast, lunch and evening meal in Part B, samples were collected just after the meal and at the following times after starting each meal: 0.5, 1 and 2 hours. Samples were also collected in Part B at 24 hours post-dose. When this results in multiple samples at the same time point, only one sample was collected. Change from Baseline was calculated by subtracting Baseline value from post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 1 (24 hours)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pico moles per Liter
Arm/Group | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally
Number analyzed (Participants) | 4 | 4
Pico moles per Liter
  C-PEPTIDE | 13.44 (226.572) | 55.83 (-507.439)
  GIP TOTAL | 2.23 (38.211) | 5.40 (-165.542)
  GLP-1 ACTIVE | 0.00 (NA) — NA indicates: The mean change from Baseline is 0.00, hence measure dispersion could not be calculated. | 0.00 (NA) — NA indicates: The mean change from Baseline is 0.00, hence measure dispersion could not be calculated.
  GLP-1 TOTAL | 0.56 (384.900) | 0.48 (66.682)
  GLUCAGON: number analyzed (Participants) | 1 | 3
  GLUCAGON | 0.94 (NA) — NA signifies measure dispersion was not calculated as only one participant was available. | 2.02 (72.451)
  INSULIN | 31.18 (223.783) | 7.19 (7682.607)
  PYY TOTAL | 3.05 (99.436) | 4.55 (181.246)

44. Secondary Outcome: Part C: Summary of Cmax of GSK1292263 and Sitagliptin When Co-administered
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (= post-breakfast), 1, 2, 4 (= pre-lunch), 6, 10 (= immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per mL
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 12 | 12 | 11 | 10 | 12 | 12
Nanograms per mL | 301.89 (20.128) | 284.59 (20.569) | 458.24 (39.382) | 378.12 (30.390) | 307.45 (31.323) | 360.91 (26.831)

45. Secondary Outcome: Part C: Summary of T-half and Tmax of GSK1292263 and Sitagliptin When Co-administered
Description: The time at which Cmax was observed was determined directly from the raw concentration-time data. The lag time before observation of drug concentrations in sample matrix determined as the time of the sample preceding the first quantifiable concentration. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (= post-breakfast), 1, 2, 4 (= pre-lunch), 6, 10 (= immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 15 | 12 | 13 | 12 | 12
Hour
  T-half, Day 14: number analyzed (Participants) | 12 | 12 | 11 | 10 | 12 | 12
  T-half, Day 14 | 7.60 [6.3 to 10.4] | 7.24 [6.2 to 9.1] | 7.38 [5.9 to 8.1] | 7.22 [4.9 to 9.1] | 7.85 [6.3 to 8.9] | 7.89 [7.1 to 9.7]
  T-max, Day 14: number analyzed (Participants) | 12 | 12 | 11 | 10 | 12 | 12
  T-max, Day 14 | 2.00 [1.0 to 4.0] | 2.00 [2.0 to 4.0] | 2.00 [1.0 to 4.0] | 2.00 [0.5 to 3.0] | 2.00 [1.0 to 4.0] | 2.00 [0.5 to 4.0]

46. Secondary Outcome: Part C: Summary of AUC0-24, AUC0-t of GSK1292263 and Sitagliptin When Co-administered
Description: The AUC0-10, AUC0-12 and AUC0-24 determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. When GSK1292263 was dosed once daily, blood samples were collected on Days 1, 13 and 14 immediately pre-dose (time 0) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-dose. When GSK1292263 was dosed BID, blood samples were collected on Days 1, 13 and 14, at immediately pre-morning dose, 1,2, 4, 6, 8, 10, 11, 12, 14, 16, 18 and 24 hours post-morning dose. For once daily and BID dosing regimens on Day 7, blood samples were collected at pre-dose (= post- breakfast), 1, 2, 4 (= pre lunch), 6, 10 (= immediately post-dinner) and 12 hours. When planned PK sampling results in multiple samples at the same time point, only one sample was collected.
Time Frame: Days 1, 7, 13 and 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms×hour per mL
Arm/Group | Part C: GSK1292263 50 mg BID | Part C: GSK1292263 150 mg BID | Part C: GSK1292263 300 mg BID | Part C: GSK1292263 600 mg Once Daily | Part C: Placebo | Part C: Sitagliptin 100 mg
Number analyzed (Participants) | 14 | 15 | 12 | 13 | 12 | 12
Nanograms×hour per mL
  AUC 0-24, Day 14: number analyzed (Participants) | 12 | 12 | 11 | 10 | 12 | 12
  AUC 0-24, Day 14 | 2701.81 (16.951) | 2585.15 (18.942) | 3338.49 (25.396) | 3012.70 (19.602) | 2437.10 (26.512) | 3027.99 (22.377)
  AUC 0-t, Day 14: number analyzed (Participants) | 12 | 12 | 11 | 10 | 12 | 12
  AUC 0-t, Day 14 | 2701.79 (16.955) | 2585.10 (18.944) | 3338.27 (25.407) | 3012.70 (19.602) | 2436.88 (26.520) | 3027.81 (22.388)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were reported throughout the study (approximately up to Week 62).
Description: ITT analysis set was used for reporting AE and SAE.
Groups:
- Part A: Placebo: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive matching placebo orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: GSK1292263 25 mg Orally: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive GSK1292263 25 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: GSK1292263 150 mg Orally: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive GSK1292263 150 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: GSK1292263 800 mg Orally: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive GSK1292263 800 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part A: Sitagliptin 100 mg Orally: In this part (Cohort 1), drug naïve T2DM participants were randomized to receive sitagliptin 100 mg orally in fasted condition. These doses were administered to the participants in an ascending sequence irrespective of the randomization order for placebo and sitagliptin. In Part A, study drug was administered 2 hours before the OGTT.
- Part C: GSK1292263 50 mg BID Orally: Participants were randomized to 14 days of dosing with GSK1292263 50 mg BID once daily. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: GSK1292263 150 mg BID Orally: Participants were randomized to 14 days of dosing with GSK1292263 150 mg BID once daily. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: GSK1292263 300 mg BID Orally: Participants were randomized to 14 days of dosing GSK1292263 300 mg BID. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: GSK1292263 600 mg Once Daily Orally: Participants were randomized to 14 days of dosing GSK1292263 600 mg once daily. In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: Placebo Orally: Participants were randomized to 14 days of dosing with matching placebo (administered BID). In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
- Part C: Sitagliptin 100 mg Once Daily Orally: Participants were randomized to 14 days of dosing with open-label sitagliptin 100 mg (dosed once daily with the morning dose of GSK1292263). In this part (Cohort 3 and Cohort 4), if Cohort 3 was dosed once daily, participants in Cohort 4 were enrolled to investigate the safety, tolerability, PK and PD of GSK1292263 when dosed in a BID regimen and vice versa. For once daily dosing, study drug was administered immediately after breakfast. For BID dosing, study drug was administered immediately after breakfast and immediately after the evening meal, but prior to the 10 hour PK sample.
Arm/Group | Part A: Placebo | Part A: GSK1292263 25 mg Orally | Part A: GSK1292263 150 mg Orally | Part A: GSK1292263 800 mg Orally | Part A: Sitagliptin 100 mg Orally | Part B: GSK1292263 800 mg Fasted Condition Orally | Part B: GSK1292263 800 mg Fed Condition Orally | Part C: GSK1292263 50 mg BID Orally | Part C: GSK1292263 150 mg BID Orally | Part C: GSK1292263 300 mg BID Orally | Part C: GSK1292263 600 mg Once Daily Orally | Part C: Placebo Orally | Part C: Sitagliptin 100 mg Once Daily Orally
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/11 | 0/13 | 0/4 | 0/4 | 0/14 | 0/16 | 0/12 | 0/14 | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/11 | 0/13 | 0/4 | 0/4 | 0/14 | 0/16 | 0/12 | 0/14 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 2/11 | 2/12 | 2/12 | 4/11 | 2/13 | 0/4 | 1/4 | 4/14 | 5/16 | 1/12 | 4/14 | 4/15 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=11) | Part A: GSK1292263 25 mg Orally (N=12) | Part A: GSK1292263 150 mg Orally (N=12) | Part A: GSK1292263 800 mg Orally (N=11) | Part A: Sitagliptin 100 mg Orally (N=13) | Part B: GSK1292263 800 mg Fasted Condition Orally (N=4) | Part B: GSK1292263 800 mg Fed Condition Orally (N=4) | Part C: GSK1292263 50 mg BID Orally (N=14) | Part C: GSK1292263 150 mg BID Orally (N=16) | Part C: GSK1292263 300 mg BID Orally (N=12) | Part C: GSK1292263 600 mg Once Daily Orally (N=14) | Part C: Placebo Orally (N=15) | Part C: Sitagliptin 100 mg Once Daily Orally (N=12)
Headache (Nervous system disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.